CLINICAL TRIAL: NCT07058584
Title: Synergistic Effects of Aerobic Exercise and Repetitive Transcranial Magnetic Stimulation on Brain Connectivity and Pain Sensitivity
Brief Title: Synergistic Effects of Aerobic Exercise and Repetitive Transcranial Magnetic Stimulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Enrico De Martino, Principal Investigator, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-20240053 - Study 2
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Aerobic Exercise; Repetitive Transcranial Magnetic Stimulation (rTMS)
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants attend two laboratory sessions scheduled one week apart, as part of a randomized, crossover study. In this design, each participant receives both conditions - an active and a sham repetitive transcranial magnetic stimulation (rTMS) intervention - in a randomized order. This within-subject crossover approach allows each participant to serve as their own control, improving statistical power and reducing the influence of inter-individual variability.
Masking Description: Randomization is applied only at the participant level: each participant is randomly assigned to start with either the active or sham condition, with the alternate condition administered in the second session. The study is single-blinded, meaning that participants are blinded to the intervention type (active vs. sham), while the investigators administering the sessions are aware of the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aerobic Exercise & rTMS (Experimental): Each session includes identical procedures, except for the type of repetitive transcranial magnetic stimulation (rTMS) administered. Participants receive active rTMS in one session and sham rTMS in the other, with the order randomized. The intervention arm includes the following procedures (not in order):
  Pain pressure threshold (PPT) assessments performed three times per session
  TMS-EEG data collection conducted at two time points per session
  30 minutes of moderate-intensity cycling on a stationary bike
  Resting-state EEG recorded twice per session
  Repetitive TMS intervention: active stimulation in one session, sham stimulation in the other
  Interventions: Device: repetitive Transcranial Magnetic Stimulation; Device: Sham repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — Repetitive transcranial magnetic stimulation (rTMS) is administered using a figure-of-eight coil from MagVenture positioned over the left primary motor cortex (M1) in an anteroposterior direction. High-frequency rTMS is delivered at 10 Hz, consisting of 100 trains of 10-second duration (3000 pulses), with 20-second inter-train intervals, at ~90% of resting motor threshold (RMT) depending on participant tolerance and TMS-EEG brain response.
Device: Sham repetitive Transcranial Magnetic Stimulation — This intervention involves high-frequency repetitive transcranial magnetic stimulation (rTMS) applied over the primary motor cortex (M1), using a figure-of-eight coil. In the sham condition, the same coil is used, but it is oriented away from the scalp at an angle that prevents effective magnetic stimulation of the brain, while still producing similar auditory and tactile sensations. This allows participants to remain blinded to the intervention type, maintaining the single-blind nature of the study. The active stimulation is delivered at 10 Hz, comprising 30 trains of 10 seconds (9900 milliseconds)(3000 pulses in total), with 20-second inter-train intervals, at ~110% of the individual's resting motor threshold (rMT). Stimulation is delivered while the participant is seated at rest, and the full rTMS protocol takes approximately 15 minutes to complete.

SUMMARY:
Participants attend two sessions, one week apart, as part of a randomized crossover study involving either an active or sham intervention. Both sessions follow identical procedures, except for the TMS intervention. Each session includes: three pain pressure threshold measurements, two TMS-EEG recordings, 30 minutes of moderate-intensity exercise on a stationary bike, and two resting-state EEG recordings. Repetitive TMS is administered as an active intervention in one session and as a sham in the other, and more.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnant or breastfeeding
* Regular use of cannabis, opioids, or other drugs
* Chronic pain (i.e., pain most days within the last three months)
* Current or previous neurologic or musculoskeletal illnesses, psychiatric diagnoses, or other ilnesses (e.g., brain or spinal cord injuries, degenerative neurological disorders, major depression, cardiovascular disease, chronic lung disease, etc.)
* Current regular use of analgesic medication or other medication which may affect the trial (including paracetamol and NSAIDs)
* Recent history of acute pain (i.e., episodic migraine attacks or pain in the lower limbs)
* Abnormally disrupted sleep in 24 hours preceding experiment
* Contraindications to TMS application (history of epilepsy, metal implants in head or jaw, etc.)
* Unable to fulfil the criteria of the "Transcranial Magnetic Stimulation Adult Safety Screen"
* Presence of implanted hearing aids or metal implants on the face, including permanent makeup or tattoos.
* Lack of ability to cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cortical connectivity | Day 1
  Global and local mean field amplitude
Cortical connectivity | Day 2
  Global and local mean field amplitude

SECONDARY OUTCOMES:
Pain Pressure Threshold | Day 1
  Pain Pressure Threshold in kPa will be measured 3 times per session using handheld algometer.
Pain Pressure Threshold | Day 2
  Pain Pressure Threshold in kPa will be measured 3 times per session using handheld algometer.
Cortical excitability | Day 1
  TMS-evoked potentials from the TMS-EEG.
Cortical excitability | Day 2
  TMS-evoked potentials from the TMS-EEG.
Borg-20 | Day 1
  Questionnaire for subjective fatique level on a scale from 6 to 20, where 6 is rest and 20 is maximal exertion. We will ask the rating at different timepoints during the 30 minutes exercise.
Borg-20 | Day 2
  Questionnaire for subjective fatique level on a scale from 6 to 20, where 6 is rest and 20 is maximal exertion. We will ask the rating at different timepoints during the 30 minutes exercise.
Pain Numerical Rating Scale (NRS) | Day 1
  The subject will be asked to rate their pain during exercise on an NRS ranging from 0 to 10 with 0 corresponding to no pain and 10 corresponding to worst imaginable pain. We will ask the rating at different timepoints during the 30 minutes exercise.
Pain Numerical Rating Scale (NRS) | Day 2
  The subject will be asked to rate their pain during exercise on an NRS ranging from 0 to 10 with 0 corresponding to no pain and 10 corresponding to worst imaginable pain. We will ask the rating at different timepoints during the 30 minutes exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico De Martino, MD, PhD, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Gistrup, Denmark